CLINICAL TRIAL: NCT06421831
Title: A Multi-center, Open Label, Single-arm, Dose Ascending Clinical Trial for Evaluation of Safety and Efficacy of Gene Therapy Drug GC101 in the Treatment of Spinal Muscular Atrophy (SMA) Type 3 Patients
Brief Title: Evaluation of Safety and Efficacy of Gene Therapy Drug in the Treatment of Spinal Muscular Atrophy (SMA) Type 3 Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GeneCradle Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JLJY-GC101-SMA-010
Record Dates: First submitted 2024-05-10; First posted 2024-05-20 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Spinal Muscular Atrophy Type 3
Keywords: SMA type 3
MeSH Terms: conditions — Spinal Muscular Atrophies of Childhood

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- single dose cohort (Experimental): 1.2x10^14 vg/person of GC101 delivered one-time intrathecally
  Interventions: Genetic: GC101

INTERVENTIONS:
Genetic: GC101 — Self-complementary AAV9 carrying a codon-optimized SMN coding sequence(coSMN1) driven by CMV enhancer and chicken β-actin promoter

SUMMARY:
The study will evaluate safety and efficacy of intrathecal delivery of GC101 gene therapy drug as a treatment of spinal muscular atrophy Type 3 (SMA 3) patients.

DETAILED DESCRIPTION:
The purpose of this trial is to evaluate safety and efficacy of gene therapy drug GC101 in SMA 3 patients. Open-label, dose-escalation clinical trials of GC101 will be conducted in multiple centers in China.

GC101 will be administrated intrathecally. Short-term safety will be evaluated in 52 weeks and enter long-term follow-up study of 5 years at will. Patients will be tested at baseline and followed up at various time points.

The primary analysis for efficacy will be assessed at 12 months after treatment with GC101 on the changes from baseline HFMSE (Hammersmith Functional Motor Scale Expanded) and RULM（Revised Upper Limb Module) scores for patients of age ≥ 6 years old.

ELIGIBILITY:
Inclusion Criteria:

* ≥2 years of age on the day of signing the informed consent form;
* Genetic and clinical diagnosis of type 3 SMA with bi-allelic deletion of SMN1 of 5qSMA;
* Hammersmith Functional Motor Scale - Expanded (HFMSE) score is between 10 and 54 at screening;
* Female patients of childbearing age who are pregnant or lactating, as well as all enrolled patients （both male and female), should take effective contraceptive measures within 6 months after the treatment;
* Patients or patient's legal guardian(s) must be able to understand the purpose and risks of the study and voluntarily provide signed and dated informed consent prior to any study-related procedures being performed.

Exclusion Criteria:

* Patient who has participated in any previous gene therapy research trials;
* Patient who has AAV9 neutralizing antibody titer ≥1:200;
* Patient who has received Nusinersen within 120 days and Risdiplam within 15 days before treatment;
* Patient who requires invasive or non-invasive ventilatory support averaging≥16 hours/day at screening;
* SMN2 copy numbers >4；
* Patient who needs nasal or gastric tube feeding for eating;
* Patient who is positive for human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen, hepatitis C antibody, or treponema pallidum antibody;
* Known allergy or hypersensitivity to prednisolone or other glucocorticosteroids or their excipients
* Severe contractures at screening that interfere with either the ability to attain/demonstrate functional measures or with the ability to receive intrathecal (IT) dosing;
* Patient who has other serious diseases, such as severe cardiovascular and cerebrovascular diseases, digestive system diseases, urinary system diseases, endocrine system diseases, hematological diseases, immune system diseases, nervous system diseases (including but not limited to epilepsy, meningitis, history of convulsions or seizures, cerebrospinal fluid circulation disorders), and mental illnesses, etc.;
* Patient with previous injuries (such as upper or lower limb fractures) or surgical operations that have not fully recovered or reached a stable state;
* Vaccination no longer than 2 weeks before treatment;
* Patient who has any other condition that, in the opinion of the investigator, makes the subject unsuitable for participation in the study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2024-05-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 52 weeks
  Frequency of treatment-related adverse events (AEs), serious adverse events (SAEs), and changes from baseline in relevant clinical laboratory tests
Change from baseline on Hammersmith Functional Motor Scale - Expanded (HFMSE) scores at Month 12 | 52 weeks
  HFMSE consists of 33 activities that can be scored one of three ways: 0 for unable to perform, 1 for performs with modification/adaptation, and 2 for performs without modification.

SECONDARY OUTCOMES:
The proportion of patients whose HFMSE improvement ≥ 3 points at Month 12 | 52 weeks
  HFMSE ≥3 points：minimal clinically important differences (MCID) were considered for the outcomes:
Change from baseline on Revised Upper Limb Module (RULM) scores at Month 12 | 52 weeks
  RULM is a 20-item evaluation of upper limb function primarily used for those with SMA who are non-ambulatory (young children through adults).

OTHER OUTCOMES:
The proportion of patients whose Clinical Global Impression (CGI) is improved at Month 12 | 52 weeks
  The Clinical Global Impressions (CGI) is a widely used assessment tool in clinical practice, particularly for evaluating the severity of a patient's illness and the effectiveness of treatments. The CGI consists of two primary components:
  CGI-Severity (CGI-S): This scale measures how ill a patient is at a given time, with scores ranging from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). It reflects the clinician's overall view of the patient's mental health status based on all available information, including symptoms, behavior, and functional impairments experienced in the past week.
  CGI-Improvement (CGI-I): This scale rates the change in the patient's condition compared to a baseline state, prior to the initiation of treatment. It uses a seven-point scale where 1 indicates "very much improved" and 7 indicates "very much worse." The CGI-I captures the overall change in the patient's clinical state since the start of treatment.
The proportion of patients whose Motor Function Measure (MFM) is improved or maintained at Month 12 | 52 weeks
  The Motor Function Measure (MFM) is a validated scale specifically designed to assess motor function in individuals with neuromuscular disorders like Spinal Muscular Atrophy (SMA). It consists of 32 items that are scored on a 4-point Likert scale, reflecting a person's maximum ability to perform tasks without assistance.
Change from baseline of Forced Vital Capacity (FVC) at Month 12 ( for patients > 6 years) | 52 weeks
Change from baseline of Forced Expiratory Volume in 1 Second (FEV1) at Month 12 ( for patients > 6 years) | 52 weeks
Change from baseline of Maximal Inspiratory Pressure (MIP) at Month 12 ( for patients > 6 years) | 52 weeks
Change from baseline of Maximal Expiratory Pressure (MEP) at Month 12 ( for patients > 6 years) | 52 weeks
Change from baseline of 6 minutes walk test (6MWT) at Month 12 (for ambulatory patients) | 52 weeks
  The 6MWT is used for ambulatory participants with SMA and measures the total distance walked in 6 minutes.
Change from baseline of SMA Independence Scale (SMAIS) at Month 12 | 52 weeks
  The SMA Independence Scale (SMAIS) is a self-reported questionnaire to assess the amount of assistance patients require to perform daily activities. Higher SMAIS scores indicate greater independence.
  (range: 0-44).

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No